CLINICAL TRIAL: NCT04825236
Title: A Feasibility Trial of the MyVoice:CF Decision Aid to Address the Reproductive Health Needs of Women With Cystic Fibrosis
Brief Title: MyVoice:CF Decision Aid for Women With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Traci Kazmerski, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20050174
Record Dates: First submitted 2021-03-19; First posted 2021-04-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis; Contraception; Physician-Patient Relations; Pregnancy Complications
Keywords: cystic fibrosis; shared decision-making; sexual and reproductive health
MeSH Terms: conditions — Cystic Fibrosis; Pregnancy Complications; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid Users (Experimental): Patients with CF who are given access to the MyVoice:CF decision aid
  Interventions: Other: MyVoice:CF
- CF Healthcare Providers (Experimental): Members of the adult CF care team who interact with patients who have used the decision aid
  Interventions: Other: MyVoice:CF

INTERVENTIONS:
Other: MyVoice:CF — Participants will be given access to MyVoice:CF, a web-based decision aid (DA). This tool includes information about fertility, genetics, parenting, pregnancy, and breastfeeding within the context of cystic fibrosis (CF). The tool includes interactive elements designed to give users the ability to assess and reflect on their own reproductive goals and experiences and promote self-efficacy to engage in shared decision-making with their CF and women's health providers.
  Upon completion of use of the decision aid, a summary sheet is generated based on the user's interaction with the tool. This summary is supplied to the provider prior to the next appointment.

SUMMARY:
This project is a single-center feasibility study of MyVoice:CF, a patient-facing, web-based decision aid.

Aim 1) Assess the acceptability, feasibility, and usability of MyVoice:CF for women with CF and multidisciplinary adult CF providers.

Aim 2) Assess the preliminary efficacy of MyVoice:CF related to patient-provider communication, shared decision-making, knowledge, and self-efficacy for women with CF related to reproductive health concerns.

DETAILED DESCRIPTION:
This study seeks to test a decision aid created to address the disease-specific reproductive health concerns of women with cystic fibrosis. The decision aid was built out of research done by studies previously approved by the University of Pittsburgh IRB. These studies determined the information and decision support needs of women with cystic fibrosis concerning their sexual and reproductive health care.

The purpose of this study is to pilot the decision aid prototype to evaluate its feasibility, appropriateness, and acceptability.

Screening for eligibility will be conducted prior to a potential participant's visit with their CF care team. Eligible patients will be contacted via phone. Interested patients will be consented and asked to schedule a time to complete the web-based decision aid in its entirety and complete a follow up qualitative interview.

The investigators will also ask participants if they are interested in two optional activities: having their screen activity on MyVoice:CF recorded for analysis and having their next appointment with their CF team recorded for conversation analyses. The RC will explain these recordings will be de-identified prior to analysis and that no one outside of the study team will see the screen capture data, listen to the recording, or read the full transcript.

Data collection: After giving consent to participate, participants will be given the link for the baseline survey, hosted on REDCap, by the RC/RA. They will also schedule a time to 1) complete the web-based decision aid and 2) complete an exit survey about the aid.

Immediately following their next visit with the CF care team, they will complete a survey to assess the tool's impact on their interaction with the team and their receipt of reproductive health care and complete a qualitative interview on the tool and its impact on their team interaction.

The subsequent 3-month and 6-month surveys will also be completed via REDCap, and participants will be given the link via email, with phone calls as necessary to prompt completion. Six months after the last recruited patient has completed their run through of the tool, the adult CF care team (n=11) will be asked to complete an anonymous survey about their experiences with patients who have used the tool. Following this, a focus group will be conducted with the care team to discuss the perceived feasibility, appropriateness, and acceptability of the tool from the provider perspective.

Data Analysis:

Descriptive statistics will summarize feasibility and acceptability data. The System Usability Scale will be assessed via the accepted scoring scale. The investigators aim for >80% use of the tool (REACH), implementation integrity (IMPLEMENTATION), and satisfaction with MyVoice:CF (MAINTENANCE). Effectiveness will be assessed by fitting generalized linear mixed models with fixed effects for "period" and random effects for cluster. For outcomes assessed longitudinally, there will be an additional random effect for subject. Assuming a conservative ICC of 0.05, 5% type I error, and 15% attrition, our anticipated sample size would yield 80% power to detect mean differences of 0.41 for any of our continuous outcomes. Reproductive health outcomes and care-seeking variables will be compared to estimates from recent survey data as well as the National Survey for Family Growth (NSFG) as a U.S. general population estimate. NSFG comparisons will be adjusted for demographic differences. Survey data will be analyzed using SAS v9.4.

Thematic analysis of interview transcripts will be conducted by research study staff and decision aid developers to identify key themes produced by the pilot testing process. Themes will be evaluated and used to refine the existing prototype and develop a finalized version of the decision making tool. Data collected from the decision aid will not be collected for research purposes and will not be analyzed; it will be used to test that the data collection system is functioning correctly.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender female
* Age 18-44 years
* English-speaking
* Diagnosed with cystic fibrosis

Exclusion Criteria:

* Men
* Women under 18 (this tool was not designed to appropriately address the sexual and reproductive health needs and experiences of the adolescent population)
* Patients who have no computer and internet access and would be unable to access the tool
* Patients who are unable to consent

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention | Patients- T2 (within 24 hours of intervention)
  Four-item measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean, with a higher score indicating higher acceptability.
Intervention Appropriateness Measure | Patients- T2 (within 24 hours of intervention)
  Four-item measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean, with a higher score indicating greater acceptability.
System Usability Scale | Patients- T2 (within 24 hours of intervention)
  Ten-item measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean, with a higher score indicating greater usability.
Perceived Value of Tool to Providers | Providers- T5 (6 months after recruitment ends)
  Five-item measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean, with a higher score indicating higher perceived value.
Acceptability of intervention to providers | Providers- T5 (6 months after recruitment ends)
  Four-item measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean, with a higher score indicating higher acceptability.
Intervention Appropriateness Measure for providers | Providers- T5 (6 months after recruitment ends)
  Four-item measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean, with a higher score indicating greater acceptability.

SECONDARY OUTCOMES:
ReproKnow (adapted) | T3 (up to 12 weeks post-tool use) compared to T0 (baseline)
  Completion of a 10-item multiple choice instrument adapted from ReproKnow, a validated instrument for assessing knowledge of reproductive health in rheumatic diseases. Answers will be coded as correct or incorrect. The percentage of correct responses across the 10 questions will be calculated for each participant. The score range is 0 to 100%. Participant knowledge will be measured at baseline and following their first clinic visit post-use of the tool to assess the sustained impact of the decision aid on knowledge.
Shared Decision-Making (collaboRATE) | T3 (up to 12 weeks post-tool use) ; T4 (up to 24 weeks post-tool use)
  Three-item measure with 5-point Likert scale questions of 0 (no effort was made) to 4 (every effort was made) to assess shared decision-making between patients and providers. The mean of all three items is calculated. Higher scores represent more shared decision-making.
Perceived Efficacy in Patient-Physician Interactions | T3 (up to 12 weeks post-tool use)
  Five-item measure with 5-point Likert scale questions from 1 (not at all confident) to 5 (very confident). Score is determined by the sum (possible range of 5 to 25) with higher score indicating higher perceived efficacy in communicating with providers
Reproductive Self Efficacy | T3 (up to 12 weeks post-tool use) compared to T0 (baseline)
  Five-item measure with 5-point Likert scale questions from 1 (not at all confident) to 5 (very confident). Score is determined by the sum (possible range of 5 to 25) with higher score indicating higher perceived efficacy in communicating with providers.
Change in Pregnancy Intention | Change between T3 (up to 12 weeks post-tool use) and T0 (baseline)
  Desire to Avoid Pregnancy scale- 14-item measure with 5-point Likert scale questions from 0 (strongly agree) to 4 (strongly disagree). Score is determined by calculating the mean (range of 0-4) with higher scores reflecting a higher desire to avoid pregnancy
Quantity and quality of reproductive conversations | T3 (up to 12 weeks post-tool use) ; T4 (up to 24 weeks post-tool use)
  Three-item measure. Did you discuss reproductive goals with your CF team- Yes/no/don't know; [if yes] Rate the quality of the discussion from 0 (very poor) to 4 (very good); [if no] why not discussed- Assessed by participant response to a multiple choice item asking why reproductive goals were not discussed (time, patient comfort, provider comfort, unfamiliar provider, other visit priorities, unsure, other)
Participant Feedback to Tool | T3 (up to 12 weeks post-tool use)
  Informed by in-depth interviews with women about their likes and dislikes of the MyVoice tool, their perceived barriers and facilitators to its use, if/how MyVoice could be used in their own lives. Questions also assess whether the CF team discussed reproductive health and if/how MyVoice influenced those decisions.
Participant Change in Contraceptive Use | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  Assessed by participant responses to a multiple choice item asking which methods of contraception they are currently using (in the past 2 weeks). Reasons for non-use assessed by response to a multiple choice item asking why they are not currently using contraception.
Participant Confidence in Contraceptive Method Selection | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  Assessed by participant responses to a 5-point Likert scale regarding satisfaction with current contraceptive method(s). Response options range from 1 ("Very Unsatisfied") to 5 ("Very Satisfied").
Participant number of pregnancies during study | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  Assessed by participant-reported survey responses to a Yes/No item about whether a pregnancy has occurred since enrollment.
Participant receipt of infertility care | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  Yes/No to question of whether pregnancy occurred with or without medical intervention; multiple choice question assessing what type of medical intervention was used.
Participant receipt of preconception counseling | T4 (up to 24 weeks post-tool use)compared to T0 (baseline)
  Y/No to question of whether pregnancy was discussed prior to conception with health care provider; multiple choice question of source of preconception care
Participant Desire for future pregnancy | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  3-item measure assessing feelings about future pregnancy- question on desire for future child, question on preferred timing, question on emotional response if she became pregnant now.
Intent to breastfeed | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  1-item measure asking how participant would feed a future baby (breastfeeding, bottle feeding, combination, unknown)
Receipt of SRH care | T4 (up to 24 weeks post-tool use) compared to T0 (baseline)
  Asks whether participant has visited a clinic for any of the following over the course of the study: birth control prescription, birth control counselling, pregnancy test, preconception counseling, prenatal care.

CONTACTS AND LOCATIONS:
Overall Officials: Traci M Kazmerski, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No